CLINICAL TRIAL: NCT05185908
Title: The Effects of Lateral 45° Downward Position and Carbon Dioxide Pneumoperitoneum on the Optic Nerve Sheath Diameter in Patients Undergoing Laparoscopic Transperitoneal Nephrectomies: A Prospective Observational Study
Brief Title: The Effects of Lateral 45° Downward Position on the Optic Nerve Sheath Diameter
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associate Professor, Istanbul University
Other Study IDs: OpticNerveSheathIU
Record Dates: First submitted 2021-12-05; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Optic Nerve Sheath Diameter
Keywords: Carbondioxide pneumoperitoneum; Optic nerve; Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: The patients undergoing laparoscopic transperitoneal nephrectomy.
  Interventions: Procedure: Measurement of the optic nerve sheath diameter by ultrasound-guidance.

INTERVENTIONS:
Procedure: Measurement of the optic nerve sheath diameter by ultrasound-guidance. — Measurement of the optic nerve sheath diameter (ONSD) by ultrasound guidance can be used in the diagnosis of increased ICP. The investigators interrogated the effects of lateral 45° downward position and CO2 insufflation on ONSD in patients undergoing laparoscopic transperitoneal nephrectomy.

SUMMARY:
Trendelenburg position and carbon dioxide (CO2) pneumoperitoneum are in association with increased intracranial pressure (ICP) reflected by the optic nerve sheath diameter (ONSD). Measurement of ONSD by ultrasound (US) guidance can be used in the diagnosis of ICP. The investigators interrogated the effects of lateral 45° downward position and CO2 insufflation on ONSD in patients undergoing laparoscopic transperitoneal nephrectomy.

DETAILED DESCRIPTION:
Transperitoneal laparoscopic nephrectomy is a popular and increasingly used alternative to the laparoscopic retroperitoneal approach because of benefits such as minimal invasion, the transperitoneal path provides a larger working space and familiar anatomic landmarks. This technique requires a steep (35° to 45°) lateral downward (SLD) position and a CO2 pneumoperitoneum. SLD may lead to pathophysiological changes such as pulmonary dysfunction with the formation of atelectasis and increasing airway pressure as well as ocular complications. These are firstly reported 2 patients with bilateral ischaemic optic neuropathy (ION) after a da Vinci robotic-assisted procedure. SLD has raised concerns that prolonged elevation of venous pressure in the head may increase the risk of developing ION. However, a few investigations have yet been made into intraoperative changes in intraocular pressure (IOP) and optic nerve sheath diameter (ONSD) - correlating with intracranial pressure (ICP) - and their adverse ocular effects. The operative conditions get better the steeper the positioning, providing an excellent intraabdominal view and probably less bleeding. The hypothesis of the study is that patients placed in SLD for several hours have a high risk for ocular changes and peri- and postoperative complications. The aim of this study was to investigate the influence of capnoperitoneum and permanent 45° SLD on IOP and ONSD in patients undergoing laparoscopic transperitoneal nephrectomy. The investigators also analyzed the hemodynamic and respiratory parameters, duration of surgery during laparoscopic nephrectomy. Perioperative and postoperative complications were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years who have undergone laparoscopic transperitoneal nephrectomy.

Exclusion Criteria:

* Those who have neurological and cerebrovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty-six patients who have undergone laparoscopic transperitoneal nephrectomy in the period of December 2016 and February 2017 were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
optic nerve sheath diameter | up to 24 hours
  Measurement of optic nerve sheath diameter by ultrasound (US) guidance can be used in the diagnosis of increased intracranial pressure (ICP).

SECONDARY OUTCOMES:
Respiratory parameters | up to 24 hours
  Peak inspiratory pressure
Hemodynamic parameters | up to 24 hours
  Mean arterial pressure

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verdonck P, Kalmar AF, Suy K, Geeraerts T, Vercauteren M, Mottrie A, De Wolf AM, Hendrickx JF. Optic nerve sheath diameter remains constant during robot assisted laparoscopic radical prostatectomy. PLoS One. 2014 Nov 4;9(11):e111916. doi: 10.1371/journal.pone.0111916. eCollection 2014. PMID 25369152
- [Background] Chin JH, Seo H, Lee EH, Lee J, Hong JH, Hwang JH, Kim YK. Sonographic optic nerve sheath diameter as a surrogate measure for intracranial pressure in anesthetized patients in the Trendelenburg position. BMC Anesthesiol. 2015 Mar 31;15:43. doi: 10.1186/s12871-015-0025-9. eCollection 2015. PMID 25861241
- [Background] Blecha S, Harth M, Schlachetzki F, Zeman F, Blecha C, Flora P, Burger M, Denzinger S, Graf BM, Helbig H, Pawlik MT. Changes in intraocular pressure and optic nerve sheath diameter in patients undergoing robotic-assisted laparoscopic prostatectomy in steep 45 degrees Trendelenburg position. BMC Anesthesiol. 2017 Mar 11;17(1):40. doi: 10.1186/s12871-017-0333-3. PMID 28284189
- [Derived] Atasever AG, Salviz EA, Senturk Ciftci H, Bingul ES, Sivrikoz N, Erdem S, Savran Karadeniz M. The Effects of Lateral 45 degrees Head-Down Position and Carbon Dioxide Pneumoperitoneum on the Optic Nerve Sheath Diameter in Patients Undergoing Laparoscopic Transperitoneal Nephrectomies: A Prospective Observational Study. J Laparoendosc Adv Surg Tech A. 2023 Feb;33(2):171-176. doi: 10.1089/lap.2022.0344. Epub 2022 Aug 25. PMID 36036829